CLINICAL TRIAL: NCT04196530
Title: Phase 1 Open-Label Dose Escalation Study of BDB001 as a Single Agent and in Combination With Atezolizumab in Subjects With Advanced Solid Tumors
Brief Title: BDB001-102: Open Label Dose Escalation of BDB001 in Combination w Atezolizumab
Acronym: EIK1001
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eikon Therapeutics (Industry)
Collaborators: Seven and Eight (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BDB001-102
Record Dates: First submitted 2019-12-10; First posted 2019-12-12 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Tumor, Solid
Keywords: TLR7/8; Immuno-oncology; EIK1001
MeSH Terms: conditions — Neoplasms | interventions — BDB001; atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Escalation of BDB001 with atezolizumab (Experimental): This part of the study will follow a traditional 3+3 dose escalation design.
  Each successive group of patients will be enrolled at an incrementally higher dosage until the Maximum Tolerable Dose (MTD) or Recommended Phase 2 Dose (RP2D) of BDB001 with atezolizumab is reached.
  Interventions: Drug: BDB001 (EIK1001); Drug: Atezolizumab
- Dose Expansion of BDB001 with atezolizumab (Experimental): At the end of the dose escalation part of the study, the BDB001 dose to be used in combination with atezolizumab in the expansion part of the study will be established after thorough review of all available safety, preliminary efficacy, PK and PD data.
  A biologically active dose will be selected that is either the MTD, if one was established in the escalation part, or an RP2D if no MTD was established. Approximately 20 additional subjects will initially be enrolled in the dose expansion part.
  Interventions: Drug: BDB001 (EIK1001); Drug: Atezolizumab

INTERVENTIONS:
Drug: BDB001 (EIK1001) — BDB001 (EIK1001) is an immunotherapy agent.
Drug: Atezolizumab — Atezolizumab is a is a fully humanized, engineered monoclonal antibody of IgG1 isotype against the protein programmed cell death-ligand 1 (PD-L1). Atezolizumab has an acceptable preclinical safety profile and is approved as an IV therapy for a variety of advanced malignancies.
  Other Names: Tecentriq

SUMMARY:
A Phase 1 Open-label Dose Escalation Study of BDB001 in Combination with Atezolizumab in Subjects with Advanced Solid Tumors

DETAILED DESCRIPTION:
This clinical trial is a study of an experimental drug called BDB001. BDB001 is a Toll-like receptor (TLR) agonist that activates the immune system.

The primary objectives of this study are to evaluate the safety and tolerability of BDB001 in combination with atezolizumab (Tecentriq) in subjects with unresectable or metastatic solid tumors who have relapsed or are refractory to standard treatment or for whom there is no approved therapy.

This is a multi-center, open-label, dose escalation/dose expansion Phase 1 study of BDB001 in combination with atezolizumab.

The study will be conducted in two separate but independent parts: a dose escalation part with BDB001 and atezolizumab and a dose expansion part of BDB001 in combination with atezolizumab.

ELIGIBILITY:
Inclusion

Participants are eligible to be included in the study only if all of the following criteria apply:

1. Be 18 years of age on day of signing informed consent
2. Subjects with histologically or cytologically confirmed advanced or metastatic solid tumors who have disease progression after treatment with all available therapies for metastatic disease that are known to confer clinical benefit, or are intolerant to treatment, or refuse standard treatment. Note: there is no limit to the number of prior treatment regimens
3. A male participant must agree to use contraception during the treatment period and for at least 120 days after the last dose of study treatment and refrain from donating sperm during this period
4. A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

   1. Not a woman of childbearing potential (WOCBP)
   2. A WOCBP who agrees to follow contraceptive guidance during the treatment period and for at least 120 days after the last dose of study treatment
   3. A highly effective method of contraception is defined as one that results in a low failure rate (i.e., less than 1% per year, when used consistently and correctly)
5. Evidence of progressive disease (PD) within 3 months of signing the informed consent form
6. Have measurable disease with at least 1 lesion meeting measurable criteria per irRECIST as assessed by the local site investigator/radiology. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions
7. Eastern Cooperative Oncology Group (ECOG) score of 0 - 2
8. Minimum life expectancy of 3 months
9. Have adequate organ function. Specimens must be collected within 10 days prior to the start of study treatment.

   * Hematological: ANC ≥1500/µL; Platelets ≥100 000/µL; Hemoglobin ≥9.0 g/dL or ≥5.6 mmol/L
   * Renal: serum creatinine ≤ 1.5 times the ULN or estimated creatinine clearance ≥ 60 mL/min (Cockcroft and Gault formula [http://www.mdcalc.com/creatinine-clearance-cockcroft-gault-equation/])
   * Hepatic: Total bilirubin ≤1.5 ×ULN or direct bilirubin ≤ULN for participants with total bilirubin levels >1.5 × ULN; AST (SGOT) and ALT (SGPT) ≤2.5 × ULN (≤5 × ULN for participants with liver metastases)
   * Prothrombin time (PT) and partial thromboplastin time (PTT) ≤ 1.5 x ULN
10. Recovery (to baseline or to Grade 1 or less) from prior treatment-related toxicities except alopecia. Participants with ≤Grade 2 neuropathy may be eligible. Note: If participant received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study treatment.
11. Ability to comply with treatment, laboratory monitoring and required clinic visits
12. The participant (or legally acceptable representative if applicable) provides written informed consent for the trial

Exclusion

Participants are excluded from the study if any of the following criteria apply:

1. A Woman of Child Bearing Potential who has a positive urine pregnancy test (e.g. within 72 hours) prior to treatment. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
2. Prior exposure to TLR 7 agonists, such as GS-9620, imiquimod, TMX 101, resiquimod, MEDI9197, and 825A, or TLR 9 agonists such as SD-101, tilsotolimod (IMO-2125), MGN1703, GNKG168, DUK-CPG-001 and CMP-001 for treatment of the solid tumor the subject is currently being evaluated for treatment with BDB001.
3. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor such as CTLA-4, OX40, and CD137, and was discontinued from that treatment due to a Grade 3 or higher irAE.
4. Received previous therapy for malignancy within 21 days prior to administration of study drug, including any investigational agents (other than BDB001), chemotherapy, immunotherapy, biological or hormonal therapy. Subjects receiving systemic interferons or IL-2 must have discontinued the drug 4 weeks or 5 half-lives (whichever is longer) prior to initiation of study treatment because these drugs could potentially increase the risk of autoimmune conditions when given in combination with atezolizumab. Subjects receiving nitrosoureas or mitomycin C must have discontinued the drug 6 weeks prior to initiation of study treatment.
5. Subjects who are receiving a RANKL inhibitor such as denosumab prior to enrollment must be willing and eligible to receive a bisphosphonate instead; denosumab could potentially alter the activity and the safety of atezolizumab.
6. Major surgery within 4 weeks of first dose of study drug
7. Has received prior radiotherapy within 2 weeks of start of study treatment. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-CNS disease
8. Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist) are live attenuated vaccines and are not allowed
9. Currently receiving medications known to be strong inhibitors of CYP1A and CYP3A and strong/moderate inducers of CYP1A and CYP3A
10. Receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug. The use of physiologic doses of corticosteroids may be approved after consultation with the Sponsor.
11. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 21 days prior to the first dose of study treatment. Note: Participants who have entered the follow-up phase of an investigational study may participate as long as it has been 21 days after the last dose of the previous investigational agent
12. History within last 6 months of New York Heart Association Class III or IV heart failure, acute myocardial infarction, angina pectoris, uncontrolled arrhythmia, acute coronary syndromes, stent placement, uncontrolled hypertension
13. QTc interval value > 470 msec (using Fridericia's Correction)
14. Left ventricular ejection fraction (LVEF) < 50% by echocardiogram (ECHO) or multigated acquisition (MUGA) scan
15. Has known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e., without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study treatment (Kim 2017). Brain MRI is preferred to document stability of existing brain metastases. If MRI is medically contraindicated, CT with contrast is an acceptable alternative.
16. Has severe hypersensitivity (≥Grade 3) to atezolizumab and/or any of its excipients
17. Has a known history of human immunodeficiency virus (HIV) infection. No HIV testing is required unless mandated by local health authority
18. Known active hepatitis A, B or C. Subjects who are HBsAg+ and have DNA load < 2000 IU/mL (104 copies/mL) are eligible to participate in the study provided they meet the ALT and bilirubin inclusion criteria.
19. Has a known additional malignancy that is progressing or has required active treatment within the past 3 years with the exception of basal cell carcinoma of the skin, squamous cell carcinoma of the skin that has undergone potentially curative therapy, in situ cervical cancer, prostate cancer that is not actively being treated, and malignancies which have been treated with curative surgery and have not recurred.
20. Has an active infection requiring systemic therapy
21. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the participant's participation for the full duration of the study, or is not in the best interest of the participant to participate, in the opinion of the treating investigator
22. Has a known psychiatric or substance abuse disorder that would interfere with the participant's ability to cooperate with the requirements of the study
23. Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of study treatment.
24. Has had an allogenic tissue/solid organ transplant
25. Active autoimmune disease that has required systemic treatment in past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed.
26. Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis
27. History of interstitial lung disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-11-21 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-08-15 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability: incidence of adverse events and any dose limiting toxicity | up to 21 months
  Safety and tolerability of BDB001 in combination with atezolizumab as measured by the incidence of adverse events and any dose limiting toxicities (DLT)
Determine Maximum Tolerated Dose (MTD) or recommended Phase 2 Dose (RP2D) | from first dose to 21 days after first dose for each patient
  Determination of the MTD or RP2D by assessing the frequency and severity of adverse events related to BDB001 when given in combination with atezolizumab using CTCAE version 5.0 to categorize adverse event severity

SECONDARY OUTCOMES:
Radiographic Determination of Tumor Response after BDB001 in combination with atezolizumab dosing | At the beginning of Cycle 3 (every cycle is 21 days) up to 30 months after the first dose for each patient
  Radiographic determination of tumor response in subjects dosed with BDB001 and atezolizumab using irRECIST

CONTACTS AND LOCATIONS:
Overall Officials: Harry Raftopoulos, MD, Study Chair — Eikon Therapeutics
Locations (5):
- United States (5):
  - Angeles Clinic, Los Angeles, California
  - Florida Cancer Specialists, Sarasota, Florida
  - Tennessee Oncology, Nashville, Tennessee
  - NEXT Oncology, San Antonio, Texas
  - South Texas Accelerated Research Therapeutics (START), San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No